CLINICAL TRIAL: NCT05472610
Title: A Phase II Clinical Study of CD19-targeted Chimeric Antigen Receptor (CAR) T Cells Injection, for Relapsed and Refractory (R/R) Large B-cell Lymphoma
Brief Title: Study of Efficacy of BZ019 in Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mengchao Cancer Hospital (Other)
Collaborators: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZ019R-A-01
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Large B-cell Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BZ019 (Experimental): The subjects are enrolled into single-dose(1～5x10^6/kg) of BZ019 ( non viral vector CD19-targeted Chimeric Antigen Receptor (CAR) T Cells Injection).
  Interventions: Biological: BZ019

INTERVENTIONS:
Biological: BZ019 — A treatment program will include lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by single-dose of BZ019 administered intravenously (IV).

SUMMARY:
This is a single arm,open-label, non-randomized phase 2 study to determine the efficacy of BZ019 in relapsed or refractory CD19+ B-cell Lymphoma subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1）Written informed consent must be obtained prior to any screening procedures;
* 2）75 ≥Age ≥ 18 years subjects；
* 3）Subjects who meet the following diagnostic and therapeutic requirements when screening: A）The diagnosis of B Cell NHL was consistent with WHO classification in 2017；

B） Subjects must be accepted adequate treatment before and have received at least 2 lines of treatment or relapse or progress after autologous hematopoietic stem cell transplantation, and the treatment history at least include:

a）Treatment by CD20 monoclonal antibody (Rituximab) except for CD20 negative; b) A chemotherapy regimen containing anthracyclines.

C）With Relapsed or refractory large B-cell lymphoma when screening:

a) The definition of relapsing is as follows：PD occurs at least after remission (including PR or CR) with standard therapy (including Rituximab) b) The definition of refractory is as follows: i) No response to the last treatment, including:The best response to the latest treatment is PD or SD; ii)Disease progression after ASCT or recurrence within ≤ 12 months (recurrence must be confirmed by biopsy), or if receiving remedial treatment after ASCT, the subject must have no reaction or recurrence after the last treatment.

D) CD19+ which was detected by immunocytochemistry or flow cytometric ;

* 4)According to the preliminary evaluation, staging and response evaluation recommendations for Hodgkin and non Hodgkin's lymphoma (2014 Edition), at least one measurable lesion was found in the screening period：the length diameter of the intranodal lesion was greater than 1.5cm,the diameter of the external lesion was greater than 1.0cm;
* 5) Life expectancy ≥12 weeks;
* 6)Baseline Eastern Cooperative Oncology Group (ECOG) score is 0 or 2 Baseline Eastern Cooperative Oncology Group (ECOG) score is 0 or 2 ;
* 7)Adequate organ function:

A)Renal function defined as:

a）A serum creatinine of ≤1.5 x ULN or Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m^2;

B）Liver function defined as:

b) Alanine Aminotransferase (ALT) ≤ 5 x ULN；Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN; c） Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air；

* 8)Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 50%, confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA)；
* 9)No blood transfusion within 1 week before signing the informed consent, sufficient bone marrow reserve is available, which is defined as: A）Absolute neutrophil count (ANC) >1x10^9/L; B）Absolute lymphocyte count (ALC) ≥ 0.5x10^9/L; C）Platelets ≥ 50x10^9/L; D）Hemoglobin > 80 g/L, for patients with bone marrow invasion, hemoglobin > 60g/L can be considered into the group;
* 10)Must have an apheresis product of non-mobilized cells accepted for manufacturing;
* 11)If the patient uses the following drugs, the following conditions should be met: A)glucocorticoids: The treatment dose of glucocorticoids must be stopped 72 hours before BZ019 infusion. However, glucocorticoids of physiological alternative dose are allowed: prednisone or its equivalent ≤ 15 mg / day; B)Immunosuppression: Any immunosuppressive medication must be stopped ≥ 4 weeks prior to enrollment; C) Antiproliferative therapies other than lymphodepleting chemotherapy within two weeks of infusion; D) Antibody use including anti-CD20 therapy within 4 weeks prior to infusion or 5 half-lives of the respected antibody, whichever is longer; E)CNS disease prophylaxis must be stopped > 1 week prior to BZ019 infusion (e.g. intrathecal methotrexate);
* 12)Women of child-bearing age and all male subjects must agree to use effective contraceptive methods until BZ019 are no longer present in the body (detected by PCR).

Exclusion Criteria:

* • Patients who have previously received any anti-CD45, anti-CD19 or anti-CD3 therapy;

  * Patients who have previously received any adoptive T cell therapy or gene therapy products, including CAR-T therapy;
  * Active Central Nervous System (CNS) involvement by malignancy or secondary CNS involvement
  * History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or self-immune disease with CNS involvement.
  * Prior allogeneic HSCT.
  * Patients with positive hepatitis B (HBsAg and / or HBcAb positive, except for those with positive surface antibody alone) or hepatitis C serological markers;
  * HIV positive or Treponema pallidum positive patients.
  * Patients with uncontrollable active or life-threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours before infusion);
  * Patients with unstable angina and / or myocardial infarction within 6 months before screening, or patients with serious or uncontrollable other diseases (such as unstable or uncompensated respiratory, heart, liver or kidney diseases) during screening;

Previous or concurrent malignancy with the following exceptions:

1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
3. A primary malignancy which has been completely resected and in complete remission for ≥ 5 years

   * Pregnant or nursing (lactating) women.
   * Patients with uncontrolled arrhythmia.
   * Patients on oral anticoagulation therapy within 1 week prior to BZ019 infusion.
   * Patients with active neurological auto immune or inflammatory disorders(e.g. Guillain Barre Syndrome, Amyptrophic Lateral Sclerosis)
   * Other conditions, such as compliance, that the investigators consider should not be included in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Month 3
  Clinical response will be assessed by RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Month 12
  Peak Plasma Concentration (Cmax)
Pharmacodynamics (PD) | Month 12
  PD of IL-2, IL-4, IL-6,IL-10, IL-15, IFN-γ, TNF-α will be analysed after CAR T cell infusion
Quality of life（QOL） | Month 12
  Quality of life will be assessed by EQ-5D health Index scale

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Y, Lin Z, Zhang F, Chen X, Yang Y, Fu X, Li Z, Sun Y, Qian Q. Rapid response in relapsed follicular lymphoma with massive chylous ascites to anti-CD19 CAR T therapy using Piggy Bac: A case report. Front Immunol. 2022 Dec 1;13:1007210. doi: 10.3389/fimmu.2022.1007210. eCollection 2022. PMID 36532014